CLINICAL TRIAL: NCT04581538
Title: Digital Support for Quality Assurance in 24-hour Caregiving at Home
Acronym: 24h-quAALity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Putz (Other)
Collaborators: NOUS Wissensmanagement GmbH (Unknown); Johanniter Österreich Ausbildung und Forschung gem. GmbH (Unknown); CARITAS Rundum zu Hause betreut (Unknown); Österreichischer Gesundheits- und Krankenpflegeverband (Unknown); ipb - Institut für Personenbetreuung (Unknown); Home-Care-Management ALEXANDER WINTER e.U. (Unknown)
Responsible Party: Sponsor-Investigator, Peter Putz, Research & Development, FH Campus Wien, University of Applied Sciences
Organization: FH Campus Wien, University of Applied Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAL01
Record Dates: First submitted 2020-09-28; First posted 2020-10-09 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Age Problem
Keywords: elderly; 24-hour home care; e-learning; digital care documentation; emergency management; active and assisted living
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Three parallel arms investigate 1) the control group, where home care is being continued as before, 2) combined effects of the e-learning platform and the networking platform, and 3) effects of the entire intervention (e-learning platform, networking platform, digital care documentation). The interventions last 12 months, with effects being investigated in two follow-ups after three and 12 months. The main one-sided alternative hypothesis, assumes a positive trend from 1 ) towards 3) in the outcomes studied. Planned contrasts are:
  1. control vs. experimental arm 3 (indicating effects of the entire experimental intervention)
  2. arm 2 vs. arm 3 (indicating whether arm 3 has additional effects as compared to arm 2)
  Planned contrasts are ignored, if the overall null hypothesis is not rejected in the ANOVA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): This arm is being provided with continued home care as it was before
- E-learning platform & networking platform (Experimental): This arm is being provided with the e-learning platform and networking platform as components of the 24-h-quAALity package
  Interventions: Device: Intervention of parallel arm 2
- Entire intervention (Experimental): This arm is being provided with the entire intervention (e-learning platform, networking platform and digital care documentation)
  Interventions: Device: Intervention of parallel arm 3

INTERVENTIONS:
Device: Intervention of parallel arm 2 — This intervention consists of the e-learning platform and the networking platform from the newly developed client-server software solution "24-h-QuAALity".
  The e-learning platform offers concise evidence-based information on common clinical patterns, as well as examples of assistance, physical activity, nutrition and daily routine provided in the caregivers' mother tongues.The caregivers use the e-learning content according to the needs of their clients and their caring skills. After completing the e-learning courses they do a test to prove their knowledge.
  The networking platform supports caregivers in communicating with other caregivers and relatives of the care receiver, with special consideration of language barriers. The caregivers use the networking platform primarily to get information or exchange it, if there are uncertainties in the care.
  Arms: E-learning platform & networking platform
Device: Intervention of parallel arm 3 — Intervention Description: This interventions represents the entire 24-h-QuAALity package consisting of the e-learning platform and networknig platform as specified under "intervention 1" and the digital care documentation from the newly developed client-server software solution "24-h-QuAALity".
  The digital care documentation aims at supporting caregivers in managing their daily tasks and facilitates exchange with other health professionals and palliative supply. The caregivers use the care documentation every day. They describe the caring and household activities they have done by their clients. The integrated emergency management empowers caregivers with lifesaving first aid skills and knowledge including an integrated voice communication and emergency call system. The emergency management system is used by caregivers when an emergency happens in which life-threatening diseases have to be managed.
  Arms: Entire intervention

SUMMARY:
Due to the demographic change, there is a growing demand for professional and institutional care, as well as the need for 24-hour home care. Care receivers range from elderly people, in need of assistance with household activities only, to those with a comprehensive need for round-the-clock care. Caregivers commute between Austria and their respective home country (mainly Slovakia, Hungary and Romania) in a two or more weeks cycle. Burdensome working conditions arise mainly due to language problems, isolated coexistence with a person affected by e.g. dementia, in combination with limited professional education and quality control.

The aim of the project is the development and evaluation of a software solution for the support and quality assurance of 24-hour home care. The application software contains:

1. an information and education portal (e-learning platform)
2. a comprehensive electronic care documentation
3. an integrated emergency management
4. links to translation pages or networking opportunities with members and relatives

DETAILED DESCRIPTION:
Due to the demographic change, there is a growing demand for professional and institutional care, as well as the need for 24-hour home care. Due to the cost-efficiency and 24-hour availability, the 24-hour home care represents a cornerstone of the care of older people and, with more than 60.000 users in Austria, it represents an important alternative to family assistance and mobile care. Care receivers range from elderly people, who only need assistance with household activities, to those with a high need for a round-the-clock care. Caregivers commute between Austria and the respective home country (mainly Slovakia, Hungary and Romania) for the care work in a two or more weeks rhythm. Burdensome working conditions arise mainly due to language problems, isolated coexistence with a person affected by e.g. dementia in combination with little to no relevant professional education and quality control.

The aim of the project is the development and evaluation of a distributed client-server software solution for the support and quality assurance of 24-hour home care. The application software contains:

1. an information and education portal (e-learning platform) with interactive learning content on common diseases and short videos on recurrent care situations in German, as well as in Slovak, Hungarian and Romanian as the most frequent languages of the caregivers.
2. a comprehensive electronic care documentation that supports quality assurance and ensures transparency between people involved.
3. an integrated emergency management, which offers caregivers the opportunity to react quickly and professionally to emergencies.
4. links to translation pages or networking opportunities with members and relatives.

By using the application software, the quality of care will be supported and further result in an increase of care quality and quality of life of the older adults cared for. Due to intense longitudinal evaluation design with more than 100 involved households facilitating 24-hour home care for a period of 12 months, the efficacy will be measured multi-dimensionally. Common surveys and structured interviews of people with cognitive impairments tend to lack sensitivity to the interventions studied. Hence, a mixed-method approach has been selected that integrates 1) investigator observations, 2) interviews with caregivers, 3) interviews with relative and 4) interviews with care receivers (where possible). Trained investigators generate reliable ratings via triangulation. Field work and analysis follows the methodology developed as Toolkit ASCOT (Adult Social Care Outcomes Toolkit 11) SCT4 (self completion survey).

ELIGIBILITY:
Inclusion Criteria:

* Household with 24-hour-care service
* Household located in the federal territory of Austria
* Caregiver able and willing to comply with all study related procedures and giving informed consent
* Age 55+ years for care receivers

Exclusion Criteria:

* Death of care receiver
* Termination of 24-hour-care, due to other reasons than death of care receiver
* Interruption of 24-hour-care for at least 8 weeks

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
ASCOT (Adult Social Care Outcome Toolkit) SCT4 value - Summary Score of eight ASCOT Domain Scores related to Care Receivers | Baseline
  Metric scale. Standardized metric score ranging from -0.17 to 1, where "0" is equivalent to dead and "1" is ideal.
ASCOT (Adult Social Care Outcome Toolkit) SCT4 value - Summary Score of eight ASCOT Domain Scores related to Care Receivers | 3 Month Follow-Up
  Metric scale. Standardized metric score ranging from -0.17 to 1, where "0" is equivalent to dead and "1" is ideal.ASCOT Domain Scores related to Care Receivers
ASCOT (Adult Social Care Outcome Toolkit) SCT4 value - Summary Score of eight ASCOT Domain Scores related to Care Receivers | 12 Month Follow-Up
  Metric scale. Standardized metric score ranging from -0.17 to 1, where "0" is equivalent to dead and "1" is ideal.ASCOT Domain Scores related to Care Receivers

SECONDARY OUTCOMES:
ASCOT (Adult Social Care Outcome Toolkit) SCT4 value - Summary Score of seven ASCOT Instrument for Caregivers Scores | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  Metric scale. Standardized metric score ranging from 0 to 1, where 1 is ideal.
Project specific self-rated satisfaction and usefulness related to electronic care documentation, professional skills and qualification, and interconnectedness and communication - Summary Score of 14 project specific questions for Caregivers | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  Metric scale. Standardized metric score ranging from 0 to 1, where 1 is ideal.
Project specific self-rated satisfaction and usefulness related to electronic care documentation, care quality and conditions, and interconnectedness and communication - Summary Score of 7 project specific questions for Relatives of Care Receivers | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  Metric scale. Standardized metric score ranging from 0 to 1, where 1 is ideal.
Project specific self-rated satisfaction and usefulness related to electronic care documentation, and interconnectedness and communication - Summary Score of 4 project specific questions for Nurses | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  Metric scale. Standardized metric score ranging from 0 to 1, where 1 is ideal.
ASCOT (Adult Social Care Outcome Toolkit) SCT4 - Domain Score for Personal Cleanliness and Comfort related to Care Receivers | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
ASCOT SCT4 - Domain Score for Food and Drink related to Care Receivers | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
ASCOT SCT4 - Domain Score for Accommodation Cleanliness and Comfort related to Care Receivers | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
ASCOT SCT4 - Domain Score for Personal Safety related to Care Receivers | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
Domain Score for Social Participation and Involvement related to Care Receivers | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
ASCOT SCT4 - Domain Score for Occupation related to Care Receivers | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
ASCOT SCT4 - Domain Score for Control over Daily Life related to Care Receivers | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
ASCOT SCT4 - Domain Score for Dignity related to Care Receivers | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
ASCOT SCT4 Instrument for Caregivers - Domain Occupation | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
ASCOT SCT4 Instrument for Caregivers - Domain Control over daily life | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
ASCOT SCT4 Instrument for Caregivers - Domain Looking after yourself | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
ASCOT SCT4 Instrument for Caregivers - Domain Personal safety | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
ASCOT SCT4 Instrument for Caregivers - Domain Participation and involvement | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
ASCOT SCT4 Instrument for Caregivers - Domain Space and time to be yourself | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs
ASCOT SCT4 Instrument for Caregivers - Domain Feeling supported and encouraged | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  4-point scale, indicating (aimed for as closely as possible): 1...ideal, 2…no needs, 3…some needs, 4...high needs

OTHER OUTCOMES:
Self-perceived health of Care Receivers as specified by the European Core Health Indicators (ECHI short list) | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  Ordinal scale. The question on self-perceived health ('How is your health in general?') refers to the respondent's own assessment of his or her health, which contains five answering categories: 1) very good, 2) good, 3) fair, 4) bad, 5) very bad.
Frequency of change of Caregivers | Metric scale. Annualized rate, recorded by investigator.
  Baseline, 3 Month Follow-Up, 12 Month Follow-Up
Geriatric Depression Scale (GDS) Geriatric Depression Scale (GDS) of Care Receivers | Baseline, 3 Month Follow-Up, 12 Month Follow-Up
  Metric scale. Standardized metric score ranging from 0 to 15, where higher scores mean a better outcome. Care receivers' GDS short form (Sheikh and Yesavage 1986). 15 questions, interviewed by investigator. Each check corresponds to one score point with a maximum count of 15.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Haslinger-Bauman, PhD, Principal Investigator — FH Campus Wien, University of Applied Sciences; Franz Werner, PhD, Study Director — FH Campus Wien, University of Applied Sciences
Locations (4):
- Austria (4):
  - Home-Care-Management ALEXANDER WINTER e.U., Breitstetten
  - CARITAS Rundum zu Hause betreut, Vienna
  - ipb - Institut für Personenbetreuung, Vienna
  - Johanniter Österreich Ausbildung und Forschung gem. GmbH, Vienna

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication, upon request
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: Researchers for non-commercial purposes

REFERENCES:
- [Derived] Haslinger-Baumann E, Putz P, Hauser C, Kupka-Klepsch E, Sturm N, Werner F. Digital support for quality assurance in 24-hour caregiving at home: a randomized controlled trial investigating the effects on quality of life and professional skills of paid 24h-caregivers. BMC Geriatr. 2023 Nov 17;23(1):750. doi: 10.1186/s12877-023-04454-4. PMID 37974112
- See also: Project description of funding organization — https://projekte.ffg.at/projekt/3076586